CLINICAL TRIAL: NCT02597751
Title: Developmental Coordination Disorder: Integrating Brain Imaging and Rehabilitation to Improve Outcomes
Brief Title: DCD Imaging-Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jill Zwicker, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H14-00397
Record Dates: First submitted 2015-10-19; First posted 2015-11-05 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Motor Skills Disorders
Keywords: DCD; Neuroimaging; Rehabilitation
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): Participants are randomized to treatment group. After the first MRI scan, participants are assessed by an independent occupational therapist (before and after intervention) and participate in 10 treatment sessions with a treating occupational therapist. Following the post-treatment assessment, participants have a second MRI scan. Twelve weeks later, participants have a third, follow-up scan.
  Interventions: Behavioral: Cognitive Orientation to Occupational Performance (CO-OP)
- Waitlist control (No Intervention): Participants are randomized to the waitlist control group. After the first MRI scan, participants "wait" for 12 weeks and then have a 2nd MRI scan. Participants then have 10 treatment sessions with an occupational therapist and are assessed by an independent occupational therapist before and after treatment. Participants then have a third MRI scan to examine brain changes associated with intervention.

INTERVENTIONS:
Behavioral: Cognitive Orientation to Occupational Performance (CO-OP) — CO-OP is a cognitive approach to solving functional motor problems (Polatajko et al., 2001b). Therapists teach children a global problem solving strategy (Goal-Plan-Do-Check) as a framework for developing specific strategies for overcoming motor problems; these strategies are determined after a dynamic performance analysis by the therapist to determine where the "breakdown" is in performing the task. Occupational therapists will see children once weekly for one hour over 10 weeks as per published protocol (Polatajko et al., 2001b), plus two assessment sessions. Children will select three functional motor goals to be addressed over the course of treatment, rating their performance and satisfaction of these goals pre- and post-intervention.
  Arms: Treatment Arm

SUMMARY:
Developmental coordination disorder (DCD) affects 5-6% of the school-age population, equating to ~400,000 children, or 1-2 students in every Canadian classroom. Children with DCD find it hard to learn motor skills and perform everyday activities, such as getting dressed, tying shoelaces, using utensils, printing, riding a bicycle, or playing sports. Researchers and clinicians do not know what causes DCD or why children with DCD struggle to learn motor skills. Using MRI, this study will increase understanding of how the brain differs in children with/without DCD and determine if rehabilitation can change the brain and improve outcomes of children with the disorder.

DETAILED DESCRIPTION:
SPECIFIC OBJECTIVES AND HYPOTHESES

The proposed study proposed is designed to test the overall hypothesis that, compared to typically-developing children, children with DCD (+/- ADHD) will show differences in brain structure and function, and that rehabilitation will be associated with brain differences that reflect improvement of motor function. The investigators will address three specific objectives:

Objective 1: To characterize structural and functional brain differences in children with DCD and typically-developing children.

Hypothesis: Compared to typically-developing children, the investigators expect that children with DCD will show smaller cerebellar volume, differences in microstructural development in motor, sensory and cerebellar pathways, decreased strength of connectivity in resting, default mode, and motor networks. Children with DCD+ADHD will show poorer function in frontal and parietal areas compared to children with DCD (Langevin et al., 2014).

Approach: The investigators will use magnetic resonance (MR) imaging and advanced MR techniques to characterize brain structure and function; the investigators will use morphometry to measure cerebral and cerebellar volumes, diffusion tensor imaging (DTI) to assess microstructural development, functional connectivity MRI to measure connectivity in different brain networks, and fMRI to explore patterns of brain activation during a mental rotation task.

Objective 2: To determine if current best-practice rehabilitation intervention induces neuroplastic changes in brain structure/function and positive outcomes in children with DCD.

Hypotheses: Compared to children in the waitlist control group, the investigators expect that children in two treatment groups (DCD and DCD+ADHD) will show: (1) strengthened functional connectivity in resting, default mode, and motor networks; (2) increased integrity of the frontal-cerebellar pathway; (3) increased gray matter volume in the dorsolateral prefrontal, motor and cerebellar cortices; and (4) improved performance and satisfaction ratings of child-chosen functional motor goals. The investigators also expect that there will be a positive association between functional improvements and changes in brain structure/function.

Approach: The investigators will measure brain changes pre- and post-intervention between children with DCD and DCD+ADHD (treatment versus waitlist control). As part of treatment, children will identify three functional motor goals as a target for intervention. The investigators will use the Canadian Occupational Performance Measure (COPM; Law et al., 2005) to measure the child's rating of their performance and satisfaction pre- and post-intervention. To supplement the COPM, the occupational therapist will videotape the child performing each of their motor goals before and after intervention, and an independent occupational therapist will use the Performance Quality Rating Scale (PQRS) to objectively measure performance and change in performance (Miller et al., 2001). As a secondary measure, the investigators will evaluate fine and gross motor skills using the Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2: Bruininks & Bruininks, 2005).

Objective 3: To determine if neuroplastic and functional changes are retained at 3-month follow-up.

Hypothesis: The investigators expect children who maintained functional gains will show increased functional connectivity in brain networks, increased integrity of the frontal-cerebellar pathway, and increased gray matter volume (as in Objective #2) compared to children who did not maintain their functional gains. If most of the children maintain their functional gains, the investigators expect improvements in brain structure and function to have remained or improved from the post-intervention scan.

Approach: MR sequences and child ratings of performance and satisfaction of their functional motor goals will be repeated in both treatment and waitlist groups.

The investigators intend to recruit 30 typically-developing children, 30 children with DCD and 30 children with DCD+ADHD.

Neuroimaging analyses will include region of interest analyses (sensory, motor, and cerebellar pathways) as well as whole brain analyses using tract-based spatial statistics.

ELIGIBILITY:
Inclusion Criteria:

* children with suspected DCD based on history and results of motor testing (MABC-2) and parent questionnaire (DCDQ) and interview
* typically developing children who score at or above 25th percentile on MABC-2

Exclusion Criteria:

* a medical condition that could explain motor problem, such as cerebral palsy, significant intellectual disability, or visual impairment
* children with ferrous metal in their body

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2014-09; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | 12 weeks
  Children will rate performance and satisfaction (10 point Likert scale) of their three motor goals
diffusion tensor imaging | 12 weeks
  fractional anisotropy and diffusivity (mean, axial, and radial)

SECONDARY OUTCOMES:
Bruininks Osteretsky Test of Motor Proficiency | 12 weeks
  standardized assessment of motor skills
Performance Quality Rating Scale | 12 weeks
  qualitative observations of movement quality
functional connectivity | 12 weeks
  spatial independent components analysis of resting state networks
functional magnetic resonance imaging | 12 weeks
  patterns of brain activation during mental rotation task
morphometry | 12 weeks
  white matter, cortical gray matter, deep gray matter, and total volumes for cerebrum and cerebellum

CONTACTS AND LOCATIONS:
Overall Officials: Jill G Zwicker, PhD, OT(C), Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Zwicker JG, Missiuna C, Boyd LA. Neural correlates of developmental coordination disorder: a review of hypotheses. J Child Neurol. 2009 Oct;24(10):1273-81. doi: 10.1177/0883073809333537. Epub 2009 Aug 17. PMID 19687388
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Brain activation of children with developmental coordination disorder is different than peers. Pediatrics. 2010 Sep;126(3):e678-86. doi: 10.1542/peds.2010-0059. Epub 2010 Aug 16. PMID 20713484
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Brain activation associated with motor skill practice in children with developmental coordination disorder: an fMRI study. Int J Dev Neurosci. 2011 Apr;29(2):145-52. doi: 10.1016/j.ijdevneu.2010.12.002. Epub 2010 Dec 8. PMID 21145385
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Developmental coordination disorder: a pilot diffusion tensor imaging study. Pediatr Neurol. 2012 Mar;46(3):162-7. doi: 10.1016/j.pediatrneurol.2011.12.007. PMID 22353291
- [Background] Langevin LM, Macmaster FP, Crawford S, Lebel C, Dewey D. Common white matter microstructure alterations in pediatric motor and attention disorders. J Pediatr. 2014 May;164(5):1157-1164.e1. doi: 10.1016/j.jpeds.2014.01.018. Epub 2014 Feb 25. PMID 24576693
- [Background] Polatajko HJ, Mandich AD, Missiuna C, Miller LT, Macnab JJ, Malloy-Miller T, Kinsella EA. Cognitive orientation to daily occupational performance (CO-OP): part III--the protocol in brief. Phys Occup Ther Pediatr. 2001;20(2-3):107-23. PMID 11345506
- [Background] Miller LT, Polatajko HJ, Missiuna C, Mandich AD, Macnab JJ. A pilot trial of a cognitive treatment for children with developmental coordination disorder. Hum Mov Sci. 2001 Mar;20(1-2):183-210. doi: 10.1016/s0167-9457(01)00034-3. PMID 11471396
- [Background] Polatajko HJ, Cantin N. Developmental coordination disorder (dyspraxia): an overview of the state of the art. Semin Pediatr Neurol. 2005 Dec;12(4):250-8. doi: 10.1016/j.spen.2005.12.007. PMID 16780296
- [Background] Smits-Engelsman BC, Blank R, van der Kaay AC, Mosterd-van der Meijs R, Vlugt-van den Brand E, Polatajko HJ, Wilson PH. Efficacy of interventions to improve motor performance in children with developmental coordination disorder: a combined systematic review and meta-analysis. Dev Med Child Neurol. 2013 Mar;55(3):229-37. doi: 10.1111/dmcn.12008. Epub 2012 Oct 29. PMID 23106530
- [Derived] Malik MA, Weber AM, Lang D, Vanderwal T, Zwicker JG. Changes in cortical grey matter volume with Cognitive Orientation to daily Occupational Performance intervention in children with developmental coordination disorder. Front Hum Neurosci. 2024 May 22;18:1316117. doi: 10.3389/fnhum.2024.1316117. eCollection 2024. PMID 38841123
- [Derived] Malik M, Weber A, Lang D, Vanderwal T, Zwicker JG. Cortical grey matter volume differences in children with developmental coordination disorder compared to typically developing children. Front Hum Neurosci. 2024 May 17;18:1276057. doi: 10.3389/fnhum.2024.1276057. eCollection 2024. PMID 38826616
- [Derived] Izadi-Najafabadi S, Gunton C, Dureno Z, Zwicker JG. Effectiveness of Cognitive Orientation to Occupational Performance intervention in improving motor skills of children with developmental coordination disorder: A randomized waitlist-control trial. Clin Rehabil. 2022 Jun;36(6):776-788. doi: 10.1177/02692155221086188. Epub 2022 Apr 24. PMID 35466705
- [Derived] Izadi-Najafabadi S, Zwicker JG. White Matter Changes With Rehabilitation in Children With Developmental Coordination Disorder: A Randomized Controlled Trial. Front Hum Neurosci. 2021 Jun 3;15:673003. doi: 10.3389/fnhum.2021.673003. eCollection 2021. PMID 34149383